CLINICAL TRIAL: NCT05632757
Title: Anticipated Patient and Caregiver Burden: Impact in People with Amyotrophic Lateral Sclerosis
Brief Title: Anticipated Patient and Caregiver Burden
Acronym: FARP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RCAPHM22_0204; ID-RCB (Other: 2022-A01748-35)
Record Dates: First submitted 2022-11-16; First posted 2022-12-01 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; caregiver; burden; depression
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psychological assessments (Experimental)
  Interventions: Behavioral: Psychological assessments

INTERVENTIONS:
Behavioral: Psychological assessments — The visit will take place during a multidisciplinary assessment in the ALS Center at the Timone Hospital, Neuromuscular Disease and ALS Department. The patient will be accompanied by his/her caregiver. During this multidisciplinary assessment, the patient is present at the hospital between 8am and 4pm. The various scales and self-questionnaires can be completed during this time. The time required to complete these scales and self-questionnaires is estimated to be about 90 minutes.

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a degenerative neurological disease that causes progressive motor disability and is life threatening within a few years. The severity of the disease, the progressive loss of autonomy that leads to dependence on family and caregivers, and the lack of effective treatment sometimes leads patients to a loss of hope and to dark thoughts. The prevalence of suicidal ideation is high, with more than one third of people with ALS experiencing it. The psychological suffering of patients is often associated with that of their caregivers. The evaluation of the patients' feeling of being a burden has rarely been addressed in previous studies in ALS on the notion of burden. In this work, the investigators wish to evaluate the patient's ideas of death by also taking into account the caregiver's burden and the patient's feeling of being a burden. They wish to better understand this difficult experience by refocusing the study on the patient himself, which has rarely been addressed in studies on ALS and the notion of burden. By working on the caregiver's burden, both from the caregiver's point of view and as perceived by the patient, the investigators hope to find avenues of intervention and define actions that could help patients and their families and improve the quality of life of the patient-caregiver couple.

ELIGIBILITY:
Inclusion Criteria (patient) :

* Patient is at least 18 years of age.
* Patient having given informed consent
* Patient with ALS who has already had at least two multidisciplinary assessments in the ALS center in Marseille with an evaluation by the clinical psychologist.
* Patient with a motor handicap of grade 3 to 5 on the Rankin score
* Patient with a primary family caregiver at home (spouse, child) willing to participate in the study
* Patient who is a beneficiary of or affiliated with a social security plan

Inclusion Criteria (caregiver) :

* Adult subject at least 18 years of age.
* Subject who has given informed consent.
* Primary family caregiver of a patient with ALS who agrees to participate in the study
* Caregiver present during hospital visits.

Exclusion Criteria (patient):

* Patients with a serious and unstable associated disease, cardiac, oncological, hepatic or renal, psychiatric (schizophrenia, bipolar)
* Autonomous patient, who does not need the help of a third party for the basic gestures of daily life (Rankin 0 to 2)
* Patient living in an institution or alone at home
* Patient with cognitive impairment that interferes with activities of daily living
* Patients with marked emotional lability (spasmodic crying) due to ALS
* Patients who have had a recent diagnosis of their disease (less than 6 months)
* Patients who are unaware of the severity of their condition
* Any condition that in the opinion of the investigator or psychologist would not be compatible with the study.

Exclusion Criteria (caregiver):

* Subjects with severe and unstable cardiac, oncological, hepatic, renal or other illnesses.
* Subject with a history of psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-06-22 (Actual); Primary Completion 2026-12-22 (Estimated); Study Completion 2027-06-22 (Estimated)

PRIMARY OUTCOMES:
Impact of the patient's sense of being a burden on the patient's suicidal ideation | Inclusion visit (month 0)
  Columbia scale (highest score meaning better outcome)

SECONDARY OUTCOMES:
Relationship between the patient's feeling of being a burden living | Inclusion visit (month 0)
  Patient's Feelings of Burden Scale (highest score meaning worst outcome)
Relationship between the patient's reasons for living | Inclusion visit (month 0)
  Patient Reasons for Living Scale (highest score meaning worst outcome)
Relationship between the patient's feeling of being a burden and the caregiver's feeling of hardship | Inclusion visit (month 0)
  Patient's sense of burden scale and Zarit Caregiver Exertion Scale
Impact of the patient's sense of burden and the caregiver's sense of hardship on the quality of life of the patient and the caregiver | Inclusion visit (month 0)
  WHOQOL-Bref (World Health Organization Quality of Life, highest score meaning better outcome)
Relationship between the patient's feeling of being a burden and the motor disability | Inclusion visit (month 0)
  Beck scale (highest score meaning worse outcome)
Relationship between the patient's feeling of being a burden and the motor disability | Inclusion visit (month 0)
  Rankin scale (highest score meaning worse outcome)
Relationship between the patient's feeling of being a burden and the motor disability | Inclusion visit (month 0)
  ALSFRS score (highest score meaning better outcome)
Relationship between the depression of patient and the caregiver | Inclusion visit (month 0)
  Beck scale (highest score meaning worse outcome)
Relationship between the depression of patient and the caregiver | Inclusion visit (month 0)
  Rankin scale (highest score meaning worse outcome)
Relationship between the depression of patient and the caregiver | Inclusion visit (month 0)
  ALSFRS score (highest score meaning better outcome)
Impact of the caregiver's feeling of hardship on the patient's reasons for living | Inclusion visit (month 0)
  Patient Reasons for Living Scale (highest score meaning worst outcome)
Impact of the caregiver's feeling of hardship on the patient's reasons for living | Inclusion visit (month 0)
  Columbia Scale (highest score meaning better outcome)
Impact of the caregiver's feeling of hardship on the patient's and suicidal ideation | Inclusion visit (month 0)
  Patient Reasons for Living Scale (highest score meaning worst outcome)
Impact of the caregiver's feeling of hardship on the patient's and suicidal ideation | Inclusion visit (month 0)
  Columbia Scale (highest score meaning better outcome)
Relationship between the caregiver's perceived distress and the patient's suicidal ideation | Inclusion visit (month 0)
  Zarit scale (highest score meaning worse outcome)
Relationship between the caregiver's perceived distress and the patient's suicidal ideation | Inclusion visit (month 0)
  Columbia Scale (highest score meaning better outcome)
Relationship between caregiver's perceived distress and the patient's cognitive assessment | Inclusion visit (month 0)
  ECAS score (Cognitif Edinburgh Cognitive and Behavioural ALS Screen) (highest score meaning better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Verschueren, Principal Investigator — AP-HM
Locations (1):
- Service Maladies neuromusculaires et SLA, Marseille, France

IPD SHARING:
Plan to Share IPD: No